CLINICAL TRIAL: NCT02166775
Title: Correlation Between Sagittal Balance of the Spine and Psychopathological Profile
Status: Terminated | Type: Observational
Why Stopped: Departure of psychologist in charge of questionnaires and scales administered to patients as part of the evaluation of primary endpoint
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5541
Record Dates: First submitted 2014-06-14; First posted 2014-06-18 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Kyphosis in Depressed or Anxious Patients; Lordosis in Patients With Manic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this trial, the correlation between the psychopathological profile and sagittal balance unexplored to date spine will be studied. Indeed, a number of patients who benefited from well-conducted surgical treatment, targeted and tailored to their pathology, respond poorly to it. The investigators wonder if there are biomechanical factors or factors of psychopathological order which might influence the effectiveness of treatment. This seems logical for the entire medical community, but it has never been demonstrated in a clinical trial.

DETAILED DESCRIPTION:
The purpose of this study is to find a global diagnostic and standardized tool , easy to use, on psychopathological factors influencing the posture of the patients lombalgia so that in this will be used to use identify upstream surgery, the patients undergoing psychiatric treatment of mood rather than surgical treatment. And thus may economise a surgical operation and its complications and the related expenses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 70 years ·
* Spine surgery outpatients with or without low back pain with radicular ·- Affiliated to a social security scheme,
* Having signed an informed consent and were informed of the results of the consultation prior to inclusion

Exclusion Criteria:

* Patients having the major diseases of the spine: deformities (scoliosis, kyphosis), tumors, fractures, inflammatory and metabolic ·
* Patients having a spinal surgery history ·
* Patients difficult to inform ( emergency ward patients, patients with difficulties in oral comprehension)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kyphosis in Depressed or Anxious Patients - Lordosis in Patients With Manic
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
sagittal balance of the spine : - kyphosis in depressed or anxious patients- lordosis in patients with manic | 2 hours
  The primary endpoint was to compare the L1S1 lordosis measured in degrees relative to L1S1 lordosis expected, i-e the pelvic tilt +/- 10 ° and analyzed in relation to anxiety scores given by the Scale Hamilton Anxiety (HAM-A), depression with the Hamilton depression Scale (HAM-D) and hypomania using the Young Mania Rating Scale (YMRS). regarding the HAM-A, greater than or equal to 17 score will be considered as indicative of anxiety. For the HAM-D greater than or equal to 13 score will be considered indicative of depression. For the YMRS, greater than or equal to 20 score will be considered as indicative of a manic syndrome. It is obvious that the higher the score, the higher the importance of the disorder will be.

SECONDARY OUTCOMES:
link between the psychopathological profile and questionnaires | 2 hours
  The secondary endpoints are finding a link between the psychopathological profile of patients using self-administered questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien SCHULLER, MD, Principal Investigator — Service de Chirurgie du Rachis, Hôpital Civil, Hôpitaux universitares de Strasbourg; Yann Philippe CHARLES, MD, Study Chair — Service de Chirurgie du Rachis, Hôpital Civil, Hôpitaux universitares de Strasbourg
Locations (1):
- Dr SCHULLER Sébastien, Service de Chirurgie Du Rachis, HUS, Strasbourg, France